CLINICAL TRIAL: NCT03313934
Title: Platelet Rich Fibrin (PRF) With Hyaluronic Acid Fillers for Tear Trough Rejuvenation
Brief Title: Platelet Rich Fibrin for Tear Trough Rejuvenation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rejuva Medical Aesthetics (Other)
Responsible Party: Principal Investigator, Alex Reivitis, Clinical Research Coordinator, Rejuva Medical Aesthetics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20171835
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Tear Trough Hollowing, Under Eye Bags
Keywords: Hyaluronic Acid Filler; Platelet Rich Fibrin (PRF); Tear Trough Filler
MeSH Terms: interventions — Restylane-L; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 10 subjects will receive treatment with hyaluronic acid fillers for tear trough rejuvenation. Each subject with have one tear trough treated with HA filler mixed with Platelet Rich Fibrin, and the other tear trough injected with HA filler mixed with saline. The subject with be blind as to which tear trough contains the PRF. This will be randomly assigned for each subject and documented by the CRC.
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject will not be aware of which tear trough has the PRF condition. Additionally, the blind observer, who is going to evaluate improvement based on before/after photos, will also be blind to to which tear trough as treated with the PRF condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic Acid Filler with Saline (Placebo Comparator): For each subject, one tear trough will be injected with hyaluronic acid filler mixed with saline. This arm will act as a control to evaluate the efficacy of PRF with hyaluronic acid.
  Interventions: Combination Product: Hyaluronic Acid Filler and Saline
- Hyaluronic Acid Filler with Platelet Rich Fibrin (PRF) (Experimental): For each subject, one tear trough will be injected with hyaluronic acid filler mixed with Platelet Rich Fibrin (PRF). This study seeks to determine the efficacy of PRF in volumization of the tear trough and improvement of skin quality. This is the experimental condition.
  Interventions: Combination Product: Hyaluronic Acid Filler and Platelet Rich Fibrin (PRF)

INTERVENTIONS:
Combination Product: Hyaluronic Acid Filler and Platelet Rich Fibrin (PRF) — The use of Restylane-L to volumize the tear trough has been well documented. Combining Restylane-L with Platelet Rich Fibrin (PRF) will be studied to evaluate if PRF enhances the volumization and skin quality of the treated areas.
  Other Names: Restylane-L
  Arms: Hyaluronic Acid Filler with Platelet Rich Fibrin (PRF)
Combination Product: Hyaluronic Acid Filler and Saline — This intervention will use saline as a control to compare with PRF when mixed with hyaluronic acid fillers. Saline will dilute the HA filler in the same way PRF will, however saline as no growth factors or properties that will enhance treatment.
  Other Names: Restylane-L
  Arms: Hyaluronic Acid Filler with Saline

SUMMARY:
The purpose of this study is to investigate the efficacy and longevity of Platelet Rich Fibrin (PRF) in combination with hyaluronic acid filler for cosmetic volume restoration of the tear troughs. This study will also evaluate visible improvement in skin texture that may be attributable to the added PRF.

DETAILED DESCRIPTION:
Background: Platelet therapy is quickly becoming an integral aspect of cosmetic treatments. Most notably, Platelet Rich Plasma (PRP) has been used topically or as an injection to stimulate collagen production and enhance the efficacy of cosmetic procedures such as fat transfer, hair loss, laser treatments, and microneedling. Harvested PRP has platelets, fibrin, and white blood cells, which contribute to wound healing, neocollagenesis, and elastogenesis. Platelet Rich Fibrin (PRF) is the next generation of PRP and contains very high concentrations white blood cells, fibrin and a small amount of mesenchymal stem cells found circulating in our bloodstreams. Due to a lack of anticoagulant in the tube, PRF becomes a gel after 15-20 minutes of being isolated. This is useful in reconstructive and aesthetic medicine, which allows it to be used for cosmetic volume restoration in addition to topical indications.

Hyaluronic acid fillers have become increasingly popular in aesthetic medicine over the past two decades. Hyaluronic acid fillers are synthesized in a variety of different ways and last anywhere from 6 to 24 months, depending on the volume and location of the face or body they are injected. Fillers under the eyes in the "tear trough" area are popular treatments to allow patients to appear more refreshed and rested. Although this is an "off label" application of injectable fillers, it is extremely popular and is performed safely in many aesthetic clinics worldwide. Given that PRF can be used to restore volume, it will be determined if PRF in combination with hyaluronic acid filler will enhance resultant volume and skin quality in the treated areas.

Objective: The purpose of this study is to investigate the efficacy and longevity of Platelet Rich Fibrin (PRF) in combination with hyaluronic acid filler for cosmetic volume restoration of the tear troughs. This study will also evaluate visible improvement in skin texture that may be attributable to the added PRF.

Hypothesis: The addition of Platelet Rich Fibrin (PRF) to hyaluronic acid fillers contribute to volume restoration of the tear trough and also improve the texture and quality of the skin in the treated area. The patient will perceive a more natural and improved result on the PRF-treated side.

ELIGIBILITY:
Inclusion Criteria:

* Males/females aged 20-80 who are experiencing moderate volume loss of the tear troughs and/or under eye bags. Eligible subjects will be in generally good health and able to provide a blood sample for treatment.

Exclusion Criteria:

* Those who fall outside of the age range 20-80 years of age, with chronic health problems including but not limited to thyroid disorders, cancer, blood disease, etc. Those who do not demonstrate volume loss of the tear troughs to the degree that warrants intervention. Conversely, those who are better suited for surgical intervention as opposed to non-surgical injections will not be eligible.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Overall Tear Trough Rejuvenation | 1 month
  Restoration of volume loss and improved skin quality of the tear troughs
Improvement of Facial Rhytids | 12 months
  Reduction in wrinkles and appearance of "crepey" skin.

CONTACTS AND LOCATIONS:
Overall Officials: Kian Karimi, MD,FACS, Principal Investigator — Rejuva Medical Aesthetics
Locations (1):
- Rejuva Medical Aesthetics, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data will be collected, organized, and summarized in a manuscript to be submitted for publication. The publication will be available for other researchers to review.